CLINICAL TRIAL: NCT05235412
Title: A Cohort Study on Milk Composition, Health Outcomes, and Feeding Practices of Chinese Mothers and Infants
Acronym: Phoenix
Status: Completed | Type: Observational
Sponsor: Danone Nutricia (Industry)
Responsible Party: Sponsor
Other Study IDs: SBB20R&32016
Record Dates: First submitted 2021-12-10; First posted 2022-02-11 (Actual); Last update posted 2025-12-05 (Actual); Status verified 2024-08

CONDITIONS: Breast Feeding; Breast Milk Expression
MeSH Terms: conditions — Breast Feeding; Breast Milk Expression

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Stool, human milk, saliva
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Chinese mothers with the intention to breastfeed, and their infants.: Observational study.
  Interventions: Other: Not applicable: Observational study without any interventions.

INTERVENTIONS:
Other: Not applicable: Observational study without any interventions. — Exposures of interest: Maternal diet and lifestyle, demographics, anthropometrics, infant's health outcomes

SUMMARY:
This is a cohort study to understand the changes of breastmilk composition in the first six months after birth of Chinese infants.

DETAILED DESCRIPTION:
The relationship of breastmilk composition, the maternal gut microbiome and lifestyle factors such as diet, feeding practices and physical activity and the infant's health and gut microbiome will be investigated in this study.

ELIGIBILITY:
Inclusion Criteria:

Mothers:

1. Generally healthy mothers with the intention to breastfeed.
2. Aged 18 years and above.
3. Written informed consent.

Infants:

1. Generally healthy term born (gestational age between 37 and 42 weeks).
2. Breastfed by their mothers, either exclusively or in combination with infant milk formula, at enrolment.
3. Chinese ethnicity of mother and father.

Exclusion Criteria:

Mothers:

1. Participation in any other studies involving investigational or marketed products concomitantly or two weeks prior to entry into the study.
2. Difficulty to follow up and/or locate (e.g. known transfer to other hospitals, residing outside the city where the study site is located, or planning to move out of the current city; incapability of mothers to comply with study protocol or investigator' s uncertainty about the willingness or ability of the mothers to understand and comply with the protocol requirements.
3. Illegal drug use.
4. Regular smoking and/ or consumption of alcoholic beverages as per investigator's judgement.
5. A BMI of <18.5 or ≥ 28 pre-pregnancy or during the first regular pregnancy check around or before 16 weeks of gestational age.
6. Acute infectious disease or neoplastic disease or any kind of weakening or debilitating conditions (with history of positive, hepatitis C virus (HCV) or HIV serological test at any time during the pregnancy).
7. Presence of mastitis, fungal infections of the nipple or areola; reactivation of herpes simplex (HSV) or varicella zoster infection in the mammary or thoracic region at the time of enrolment.
8. Presence of chronic diseases such as endocrine, cardiovascular, renal, respiratory or hepatic diseases.
9. Presence of psychosis and severe post-partum depression.
10. Presence of autoimmune disease such as systemic lupus erythematosus, systemic scleroderma, ulcerative colitis, Crohn's disease, celiac disease.
11. Women whose health condition, according to the investigator's judgement, could interfere with the study conduction and assessment.
12. Mothers who have given birth to twins or multiples or infant conceived with Assisted Reproductive Technology (ART).

Infants:

1. Participation in any other studies involving investigational or marketed products concomitantly or two weeks prior to entry into the study.
2. At enrolment, any congenital abnormality, chromosomal disorder or severe disease which could interfere with the study conduct and assessment.
3. Consumption of food other than breast milk or infant formula.
4. Fully formula fed at enrolment.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Generally healthy mothers with the intention to breastfeed, and their infants.
Sampling Method: Probability Sample
Enrollment: 769 (Actual)
Dates: Start 2021-11-19 (Actual); Primary Completion 2025-07-31 (Actual); Study Completion 2025-07-31 (Actual)

PRIMARY OUTCOMES:
Changes in human milk protein concentration | Human milk samples collected at 1 month, 3 month, 6 months, 12 months, 2 years after infant birth
  Protein concentration in g/l of human milk will be analyzed
Changes in human milk fat concentration | Human milk samples collected at 1 month, 3 month, 6 months, 12 months, 2 years after infant birth
  Fat concentration in g/l of human milk will be analyzed
Changes in human milk carbohydrate concentration | Human milk samples collected at 1 month, 3 month, 6 months, 12 months, 2 years after infant birth
  Carbohydrate concentration in g/l of human milk will be analyzed
Changes in human milk energy content | Human milk samples collected at 1 month, 3 month, 6 months, 12 months, 2 years after infant birth
  Energy content in kCal/l of human milk will be analyzed
Changes in infant length | Anthropometrics collected at birth, and 1 month, 3 month, 6 months, 12 months, 2 years after infant birth
  Length measured in cm
Changes in infant head circumference | Anthropometrics collected at birth, and 1 month, 3 month, 6 months, 12 months, 2 years after infant birth
  Head circumference measured in cm
Changes in infant weight | Anthropometrics collected at birth, and 1 month, 3 month, 6 months, 12 months, 2 years after infant birth
  Weight measured in grams

SECONDARY OUTCOMES:
Variations in human milk microbiome | Human milk samples collected at 1 month, 3 month, 6 months, 12 months, 2 years after infant birth
  Analyzed by sequencing
Variations in human milk micronutrients | Human milk samples collected at 1 month, 3 month, 6 months, 12 months, 2 years after infant birth
  Analyzed by mass spectrometry
Variations in human milk oligosaccharides (HMOs) | Human milk samples collected at 1 month, 3 month, 6 months, 12 months, 2 years after infant birth
  Analyzed by mass spectrometry
Variations in human milk lipid composition | Human milk samples collected at 1 month, 3 month, 6 months, 12 months, 2 years after infant birth
  Analyzed by mass spectrometry
Variations in human milk amino acids and proteins | Human milk samples collected at 1 month, 3 month, 6 months, 12 months, 2 years after infant birth
  Analyzed by mass spectrometry
Variations in infant fecal microbiome | Infant fecal samples collected at 1 month, 3 month, 6 months, 12 months, 2 years after infant birth
  Analyzed by sequencing
Variations in maternal fecal microbiome | Maternal fecal samples collected at 1 month, 3 month, 6 months, 12 months after infant birth
  Analyzed by sequencing
Changes in infant stool consistency and frequency | Data collected at 1 month, 3 month, 6 months, 12 months after infant birth
  Data will be collected via diaries using the Brussel Infant and Toddler Stool Scale
Changes in infant feeding practices | Data collected at 1 month, 3 month, 6 months, 12 months,2 years after infant birth
  Dietary data will be collected via questionnaires
Changes in maternal body mass index | Data collected at 1 month, 3 month, 6 months, 12 months 2 years after infant birth
  Maternal weight and height will be combined to determine body mass index [kg/m2]

CONTACTS AND LOCATIONS:
Overall Officials: Jieshu Wu, Ph.D, Principal Investigator — Nanjing Medical University Jiangning Campus
Locations (1):
- Nanjing Medical University Jiangning Campus, Nanjing, Jiangsu, China

IPD SHARING:
Plan to Share IPD: No